CLINICAL TRIAL: NCT04421404
Title: A Randomized Controlled Adaptive Study Comparing COVID-19 Convalescent Plasma (CCP) to Non-immune Plasma to Limit Coronavirus-associated Complications in Hospitalized Patients
Brief Title: Effects of COVID-19 Convalescent Plasma (CCP) on Coronavirus-associated Complications in Hospitalized Patients
Acronym: CAPRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Priscilla Hsue, MD (Other)
Collaborators: Vitalant Research Institute (Other); San Francisco General Hospital (Other)
Responsible Party: Sponsor-Investigator, Priscilla Hsue, MD, Professor of Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-30794
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Results first posted 2021-08-25 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: COVID-19; Sars-CoV2
Keywords: COVID-19; Sars-CoV2; Convalescent plasma
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: Subjects enrolled in the study will be randomized using a web based randomization procedure to receive convalescent plasma versus non-immune plasma at a 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study investigators analyzing the data and participants will be blinded to the randomization. It may not be feasible to blind nursing staff to the treatment assignment to ensure proper ABO checking of the plasma unit at bedside per standard transfusion procedures, but every effort will be made to preserve blinding of the investigators, participant, and primary team providing care. An unblinded research assistant who is not involved in other aspects of the study will randomize the participant once enrolled. Randomization will be provided to an unblinded provider who is not part of the care team who will place the order for the plasma (CCP vs. control plasma) using a paper order that will not be part of the electronic medical record. The safety monitoring committee (SMC) will review study data, including unblinded data, to evaluate the safety, efficacy, study progress, and conduct of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COVID-19 Convalescent Plasma (Experimental): Subjects in the COVID-19 convalescent plasma group will receive a single infusion of 250 ml anti-SARS-CoV-2 convalescent fresh frozen plasma, ABO compatible with the patient, within 24 hours of randomization.
  Interventions: Biological: COVID-19 Convalescent Plasma (CCP)
- Placebo (Placebo Comparator): Subjects in the placebo group will receive a single infusion of 250 ml of standard fresh frozen plasma, ABO compatible with the patient, within 24 hours of randomization.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: COVID-19 Convalescent Plasma (CCP) — COVID-19 Convalescent Plasma (CCP) is a form of passive antibody therapy that involves the administration of anti-SARS-CoV-2 antibodies to a susceptible individual for the purpose of preventing or treating the infectious disease it causes. Convalescent plasma for this trial will be obtained from Vitalant (or American Red Cross if necessary). Patients identified as having recovered from COVID-19 will serve as potential donors. Potential donors will be screened using an anti-SARS-CoV-2 serologic assay and antibody levels will be determined.
  Arms: COVID-19 Convalescent Plasma
Biological: Placebo — Standard plasma will be obtained from Vitalant (or American Red Cross if necessary) and will be either collected prior to 12/1/2019 or tested and confirmed to be negative for anti-SARS-CoV-2.
  Arms: Placebo

SUMMARY:
The purpose of this study assess the efficacy and safety of anti-SARS-CoV-2 convalescent plasma in hospitalized patients with acute respiratory symptoms up to 14 days after the onset of initial symptoms.

DETAILED DESCRIPTION:
A total of 50 eligible subjects will be randomized in a 1:1 ratio to receive either convalescent fresh frozen plasma (frozen within 8 hours of collection) of PF24 (frozen within 24 hours) from blood donors who have recovered from COVID-19 containing antibodies to SARS-CoV-2 or control (standard fresh frozen plasma collected prior to 12/1/2019 or with documented negative SARS-CoV-2 antibody). Should additional anti-COVID agents (anti-viral and/or anti-inflammatory) become available for use as standard of care during implementation, the sample size will be recalculated and increased to account for the estimated impact that these agents may have on the reducing the progression to the primary endpoint of severe hypoxemia.

ELIGIBILITY:
Inclusion Criteria for Enrollment:

1. Patients ≥18 years of age
2. Hospitalized with COVID-19
3. Enrolled within 72 hours of hospitalization OR within day 14 from first signs of illness
4. Pulmonary infiltrates on chest imaging
5. Oxygenation of <95% on room air
6. Laboratory confirmed COVID-19

Exclusion Criteria

1. Contraindication to transfusion due to inability to tolerate additional fluid, such as due to decompensated congestive heart failure
2. Baseline requirement for oxygen supplementation prior to COVID-19 infection or use of positive pressure therapy for sleep disordered breathing
3. Currently experiencing severe hypoxemic failure, as defined in study endpoints
4. Prior receipt of plasma products, IVIG, or hyperimmune globulin within past 3 months
5. Not currently enrolled another interventional clinical trial of COVID-19 treatment.

Note: If taking medications with potential anti-COVID activity for the purpose of COVID-19 treatment that do not yet have data to support efficacy, such as IL-6 antagonists, these medications must be stopped prior to enrollment. Receipt of current standard of care COVID-19 treatment, including remdesivir and dexamethasone is permitted and should be recorded as a concomitant medication.

Note: Pregnancy is not exclusionary but will merit additional discussion of risks & benefits in the context of ongoing pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Hsue, MD, Principal Investigator — University of California, San Francisco; Annie Leutkemeyer, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - San Francisco General Hospital, San Francisco, California
  - UCSF Medical Center at Mount Zion, San Francisco, California
  - University of California, San Francisco Medical Center (Parnassus Campus), San Francisco, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COVID-19 Convalescent Plasma | Placebo
Started | 16 | 18
Completed (Completion of study defined as completing 29 day follow up (or died prior to day 29)) | 16 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COVID-19 Convalescent Plasma | Placebo | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [40 to 64] | 62 [49 to 74] | 57 [44 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 6 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 9 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Ventilation or Death Endpoint
Description: Number of participants that progressed to mechanical ventilation or death within the first 14 days of enrollment.
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Convalescent Plasma | Placebo
Number analyzed (Participants) | 16 | 18
Participants | 2 | 0

2. Secondary Outcome: Mechanical Ventilation or Death Endpoint
Description: Progression to mechanical ventilation or death within the first 28 days of enrollment.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Convalescent Plasma | Placebo
Number analyzed (Participants) | 16 | 18
Participants | 2 | 0

3. Secondary Outcome: 8-Point Ordinal Scale Endpoint
Description: Clinical efficacy of CCP relative to the control arm in adults hospitalized with COVID-19 according to clinical status as assessed by 8-point ordinal scale.
  8 Point WHO Ordinal Scale of Clinical Status:
  Uninfected (No clinical or virological evidence of infection) - 0
  Ambulatory (No limitation of activities) - 1 Ambulatory (Limitation of Activities) - 2
  Hospitalized Mild Disease (Hospitalized, no oxygen therapy) - 3 Hospitalized Mild Disease (Oxygen by mask or nasal prongs) - 4
  Hospitalized Severe Disease (Non-invasive ventilation or high flow oxygen) - 5 Hospitalized Severe Disease (Intubation and mechanical ventilation) - 6 Hospitalized Severe Disease (Ventilation + Additional organ support (pressors, RRT, ECMO)) - 7
  Dead (Death) - 8
Time Frame: Day 29
Population: The number of participants in the table below differs, as these are the number of participants per visit day. The number of participants decreased over the visit days as there was loss to follow up.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | COVID-19 Convalescent Plasma | Placebo
Number analyzed (Participants) | 14 | 15
score on a scale
  Day 1 | 2.43 [1 to 4] | 1.93 [1 to 3]
  Day 2: number analyzed (Participants) | 13 | 14
  Day 2 | 2.15 [1 to 4] | 2.14 [1 to 3.75]
  Day 3: number analyzed (Participants) | 12 | 13
  Day 3 | 3.92 [3 to 4] | 4 [4 to 4]
  Day 4: number analyzed (Participants) | 12 | 13
  Day 4 | 3.42 [3 to 4] | 3.69 [3.5 to 4]
  Day 5: number analyzed (Participants) | 12 | 12
  Day 5 | 2.83 [1 to 4] | 2.92 [2.5 to 4]
  Day 6: number analyzed (Participants) | 11 | 11
  Day 6 | 2.18 [0.5 to 3.5] | 2.45 [0 to 4]
  Day 7: number analyzed (Participants) | 5 | 8
  Day 7 | 3.4 [1 to 5] | 3.5 [3 to 4]
  Day 8: number analyzed (Participants) | 3 | 7
  Day 8 | 5 [4.5 to 5.5] | 2.57 [2 to 3.5]
  Day 9: number analyzed (Participants) | 3 | 7
  Day 9 | 4.67 [4 to 5.5] | 1.86 [0.5 to 3]
  Day 10: number analyzed (Participants) | 3 | 5
  Day 10 | 3.67 [2.5 to 5.5] | 1.8 [0 to 3]
  Day 11: number analyzed (Participants) | 2 | 2
  Day 11 | 5 [4.5 to 5.5] | 2.5 [2.25 to 2.75]
  Day 12: number analyzed (Participants) | 2 | 2
  Day 12 | 5 [4.5 to 5.5] | 2 [1.5 to 2.5]
  Day 13: number analyzed (Participants) | 3 | 2
  Day 13 | 3 [1.5 to 4.5] | 2.5 [2.25 to 2.75]
  Day 14: number analyzed (Participants) | 3 | 1
  Day 14 | 2 [0 to 3] | 0 [0 to 0]
  Day 15: number analyzed (Participants) | 1 | 1
  Day 15 | 6 [6 to 6] | 0 [0 to 0]
  Day 16: number analyzed (Participants) | 1 | 1
  Day 16 | 6 [6 to 6] | 8 [8 to 8]
  Day 17: number analyzed (Participants) | 1 | 1
  Day 17 | 6 [6 to 6] | 8 [8 to 8]
  Day 18: number analyzed (Participants) | 1 | 1
  Day 18 | 6 [6 to 6] | 8 [8 to 8]
  Day 19: number analyzed (Participants) | 1 | 0
  Day 19 | 6 [6 to 6] |
  Day 20: number analyzed (Participants) | 1 | 0
  Day 20 | 6 [6 to 6] |
  Day 21: number analyzed (Participants) | 1 | 0
  Day 21 | 8 [8 to 8] |
  Day 22: number analyzed (Participants) | 1 | 0
  Day 22 | 8 [8 to 8] |
  Day 29: number analyzed (Participants) | 0 | 1
  Day 29 |  | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | COVID-19 Convalescent Plasma | Placebo
All-Cause Mortality (participants affected / at risk) | 1/16 | 1/18
Serious Adverse Events (participants affected / at risk) | 2/16 | 1/18
Other Adverse Events (participants affected / at risk) | 2/16 | 1/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | COVID-19 Convalescent Plasma (N=16) | Placebo (N=18)
Intubation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Death (General disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | COVID-19 Convalescent Plasma (N=16) | Placebo (N=18)
Hypotension (transfusion reaction) (Cardiac disorders) | 0 | 1
Elevated LFTs (Hepatobiliary disorders) | 1 | 0
UTI (Infections and infestations) | 1 | 0
Elevated triglycerides (Endocrine disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was limited by the small sample of hospitalized, hypoxic patients, limiting the generalizability of the results. Most participants were beyond 72 hours of symptom onset, the period when studies suggest CCP is most likely to be beneficial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT04421404/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT04421404/ICF_001.pdf